CLINICAL TRIAL: NCT01660412
Title: Does Alkalinization of Technetium-99m Sulfur Colloid Reduce Perceived Pain Levels During Non-breast Sentinel Lymphoscintigraphy?
Brief Title: Does Alkalinization Reduce Perceived Pain Levels During Sentinel Lymph Node Imaging?
Acronym: buffering SLN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: Howard J Barnhard, Resident Research Endowment. (Unknown); UAMS DEPT of Radiology. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 31337
Record Dates: First submitted 2012-08-03; First posted 2012-08-08 (Estimated); Results first posted 2017-11-20 (Actual); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Pain
Keywords: Pain; Alkalinization; Technetium 99m Sulfur Colloid; sentinel lymphoscintigraphy?
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pH altered first (Active Comparator): The first injection administered will be the pH altered solution. The second injection will be the standard of care solution (opposite order). The remaining injections will be randomly assigned as either standard of care or pH altered.
  Interventions: Drug: ph Altered first
- Standard of Care first (Active Comparator): The first injection administered will be the standard of care solution (SOC). The second injection will be the pH altered solution. The remaining injections will be randomly assigned as either standard of care or pH altered.
  Interventions: Drug: Standard of Care First

INTERVENTIONS:
Drug: Standard of Care First — For the second injection, and randomly after that, Sodium Bicarbonate will be compounded with Tc-99m SC, to raise the pH up to ~7.40.
  Other Names: Sodium Bicarbonate second
  Arms: Standard of Care first
Drug: ph Altered first — For the first injection, Sodium Bicarbonate will be compounded with Tc-99m SC, to raise the pH up to ~7.40. For the second injection, the standard of care will be given, and randomly after that either standard of care, or pH altered will be given.
  Other Names: Sodium Bicarbonate first
  Arms: pH altered first

SUMMARY:
Pain during nuclear medicine breast lymphnode detection procedures has been reported as high as 8.8/10. Using Sodium Bicarbonate to alkalinize the radio-pharmaceutical injection, pain can safely be reduced from 6.6/10 to 4.7/10, during breast lymph node detection procedures.

In sites other then the breast, using Bicarbonate to make the injection's pH closer to natural, attempts to lower the pain levels will be performed.

Hypothesis: The perceived pain level during non breast sentinel lymph node techniques can be reduced by raising the pH of the injectate (Tc-99m SC) to near the physiologic level of pH 7.40.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting for SLN imaging for melanoma or who have had an excisional biopsy for melanoma of the thorax and appendicular structures;
* Patients scheduled to receive two or more injections of Tc-99m SC for the purpose of clinical management of melanoma or who have had an excisional biopsy for melanoma of the thorax and appendicular structures.

Exclusion Criteria:

* Patients presenting for SLN imaging of lesions involving the breast, ear, nose, and genitourinary regions;
* Patients scheduled to receive only a single injection of Tc-99m SC;
* Pregnant or breast feeding women.

Ages: 18 Years to 122 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2012-08-01 (Actual); Primary Completion 2016-12-30 (Actual); Study Completion 2016-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James A Ntambi, MD, Principal Investigator — UAMS
Locations (1):
- UAMS, Little Rock, Arkansas, United States

REFERENCES:
- [Background] Fetzer S, Holmes S. Relieving the pain of sentinel lymph node biopsy tracer injection. Clin J Oncol Nurs. 2008 Aug;12(4):668-70. doi: 10.1188/08.CJON.668-670. PMID 18676334
- [Background] Stojadinovic A, Peoples GE, Jurgens JS, Howard RS, Schuyler B, Kwon KH, Henry LR, Shriver CD, Buckenmaier CC. Standard versus pH-adjusted and lidocaine supplemented radiocolloid for patients undergoing sentinel-lymph-node mapping and biopsy for early breast cancer (PASSION-P trial): a double-blind, randomised controlled trial. Lancet Oncol. 2009 Sep;10(9):849-54. doi: 10.1016/S1470-2045(09)70194-9. Epub 2009 Aug 5. PMID 19664956
- [Result] Johnston MJ, Ntambi JA, Hilliard N, Spencer HJ, Vaughn R, Owens SS, Myrick RS, Parker LD, Garner DA, Yarbrough TL. Reducing perceived pain levels during nonbreast lymphoscintigraphy. Clin Nucl Med. 2015 Dec;40(12):945-9. doi: 10.1097/RLU.0000000000000905. PMID 26222533

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Each Participant received four injections. We tested four different injection sites. Each participant received all four injections at one site.
Period: Overall Study
Arm/Group | pH Altered First | Standard of Care First
Started | 29 | 31
Head | 1 | 4
Thorax (Including neck and buttocks) | 9 | 9
Appendicular Structures (including shoulder to wrist, back of hand, and hip to ankle) | 17 | 11
Other (Remainder of the hand and feet) | 2 | 4
Injection 1 | 29 | 31
Injection 2 | 29 | 31
Injection 3 | 29 | 31
Injection 4 | 29 | 31
Completed | 29 | 28
Not Completed | 0 | 3
Not completed — Protocol Violation | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Subjects were randomized into 1 of 2 sequence groups (A and B):
  Sequence group A. The first injection administered was the standard-of-care (SOC) solution followed by the pH-altered solution. The remaining injections were randomly assigned as either SOC solution or pH-altered.
  Sequence group B. The first injection administered was the pHaltered solution followed by the SOC solution. The remaining injections were randomly assigned as either SOC solution or pH-altered.
Arm/Group | All Study Participants
Number analyzed (Participants) | 57
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (13.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 31
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 57
Weight [Mean (Standard Deviation); unit: lbs] | 159.9 (46.1)

OUTCOME MEASURES:

1. Primary Outcome: Perceived Pain Level
Description: Immediately after receiving an injection, subjects will rate their perceived pain level, using a validated measure. Subject was asked to quantify the pain of every injection using a validated scale from 0 through 10, with 0 being no pain and 10 being severe pain that is disabling. The effect of treatment was estimated by taking the difference of the mean buffered and SOC pain scores and a paired t-test was used to test whether the mean difference was significantly different from 0. Perceived pain levels assessed after each injection were averaged for each participant.
Time Frame: immediately after administration (<1 min) of each injection (up to total 5 minutes)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Standard of Care Injection: Approximately 1mc 99mTc-SC
- PH Altered Injection: a diluted bicarbonate solution in a drop wise manner to raise the pH of the 99mTc-SC to a pH of 7.40 ± 0.05, dose Approximately 1mc
Arm/Group | Standard of Care Injection | PH Altered Injection
Number analyzed (Participants) | 57 | 57
units on a scale | 5.81 (2.24) | 4.39 (2.45)
Statistical Analysis 1: Comparison: Standard of Care Injection vs PH Altered Injection; Test type: Other; p < 0.0001, t-test, 2 sided; Mean Difference (Final Values) = 1.42, 95% CI 2-sided [0.85 to 2.00], Standard Deviation 2.17

ADVERSE EVENTS:
Time Frame: Adverse events were monitored for each injection up to 5 minutes.
Arm/Group | Standard of Care Injection | PH Altered Injection
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 11/60 | 0/60
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard of Care Injection (N=60) | PH Altered Injection (N=60)
Injection Site Pain (General disorders) | 11 | 0 — Injection site pain of 8 of 10 or less was not considered an adverse event. Injection site pain of 9/10 or 10/10 was considered an adverse event.

LIMITATIONS AND CAVEATS:
a sample size of 60 may be inadequate to generalize to all practices.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-01-17): https://cdn.clinicaltrials.gov/large-docs/12/NCT01660412/Prot_SAP_000.pdf